CLINICAL TRIAL: NCT03050944
Title: Association of the Mediterranean Diet With Fertility Outcomes: a Study Among Couples Undergoing in Vitro Fertilization Treatment
Brief Title: Association of the Mediterranean Diet With Fertility Outcomes
Acronym: MedDietIVF
Status: Completed | Type: Observational
Sponsor: Harokopio University (Other)
Collaborators: Embryogenesis Assisted Conception Unit (Unknown)
Responsible Party: Principal Investigator, Nikos Yiannakouris, Assοciate Professor of Physiology, Harokopio University, Harokopio University
Other Study IDs: 57
Record Dates: First submitted 2017-02-03; First posted 2017-02-13 (Actual); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Infertility
Keywords: Fertility; Infertility; Dietary Patterns; Mediterranean diet; Adiponectin; Follistatin; Assisted Reproduction; In Vitro Fertilization; Semen quality; Diet; IVF
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, follicular fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Lifestyle behaviour and dietary habits assessment in couples achieving pregnancy after in vitro fertilization process.
  Interventions: Other: Lifestyle behaviour and dietary habits assessment
- Controls: Lifestyle behaviour and dietary habits assessment in couples failed to achieve pregnancy after in vitro fertilization process.
  Interventions: Other: Lifestyle behaviour and dietary habits assessment

INTERVENTIONS:
Other: Lifestyle behaviour and dietary habits assessment — Lifestyle behaviour and dietary habits assessment

SUMMARY:
Infertility affects one of every six couples and one out of ten couples may seek fertility treatment such as ovulation induction and assisted reproductive technologies. With respect to diet, several dietary factors, i.e. micro-, macro-nutrients and individual food groups, have been associated with the risk of subfertility; however, more information is needed on the role of dietary factors in reproductive functions. However, evidence concerning the association between dietary patterns, such as the Mediterranean diet (MD) pattern, and fertility is scarce. The aim of this study is to investigate the relationship between preconception dietary patterns, especially the MD pattern, and in vitro fertilization (IVF) outcomes, as well as adiponectin and follistatin concentrations in the plasma and follicular fluid of women undergoing IVF treatment. Blood and follicular fluid adiponectin and follistatin concentrations will be measured on each day of the ovarian stimulation protocol. Main IVF treatment outcomes are fertilization rate, oocyte and embryo quality, implantation, clinical pregnancy and live birth rates.

DETAILED DESCRIPTION:
Infertility affects one of every six couples and one out of ten couples may seek fertility treatment such as ovulation induction and assisted reproductive technologies. There are multiple causes of infertility, including ovulatory disorders, endometriosis and sperm factors, or even psychological problems, among others. Modifiable lifestyle factors, such as diet, smoking and physical activity, may also affect fertility. With respect to diet, several dietary factors, i.e. micro-, macro-nutrients and individual food groups, have been associated with the risk of subfertility; however, more information is needed on the role of dietary factors in reproductive functions. A more comprehensive approach to investigate the associations between dietary factors and health outcomes is to assess the impact of the overall diet rather than separate foods or nutrients. However, evidence concerning the association between dietary patterns, such as the Mediterranean diet (MD) pattern, and fertility is scarce. The benefits of the MD on health have been well-publicized; it is associated with a significant reduction of overall mortality, cardiovascular disease and cancer. Adherence to the MD also seems to reduce the risk of weight gain and diabetes, conditions that raise insulin resistance and may thus lead to ovulatory infertility. Recently, adherence to MD was also associated with an increase in circulating adiponectin levels, a hormone produced by the adipose tissue that acts to reduce insulin resistance. Interestingly, adiponectin has been shown to exert actions in the female reproductive system, including the hypothalamic-pituitary ovarian axis and endometrium, and thus, it can be hypothesized that MD may exert a beneficial effect on reproductive functions through a raising effect on adiponectin levels. The aim of this study is to investigate the relationship between preconception dietary patterns, especially the MD pattern, and in vitro fertilization (IVF) outcomes, as well as adiponectin and follistatin concentrations in the plasma and follicular fluid of women undergoing IVF treatment.

Two-hundred subfertile couples undergoing IVF treatment at a Fertility Clinic in Athens (www.embryogenesis.gr/) will be invited to participate. Participants will fill out the following questionnaires: a general questionnaire to record the baseline characteristics of the subjects (age, educational level, annual income, medical history, body mass index, smoking, etc), a semi-quantitative 77-item food frequency questionnaire to assess habitual dietary intakes, and a 40-item state-trait anxiety inventory instrument to measure anxiety symptoms. Dietary patterns will be evaluated using principal component analysis and factor analysis. Adherence to the MD will be assessed with a MD-score that incorporates the inherent characteristics of this traditional diet, that is, high intake of plant foods and olive oil, low intake of meat and dairy products, and moderate intake of alcohol. Blood and follicular fluid adiponectin and follistatin concentrations will be measured on each day of the ovarian stimulation protocol. Main IVF treatment outcomes are fertilization rate, embryo quality, implantation, clinical pregnancy and live birth.

Associations between dietary patterns, adiponectin and follistatin concentrations and the IVF treatment outcomes will be tested using linear and logistic regression analyses, adjusting for potential confounders (e.g. age, smoking, anxiety symptoms, etc). The findings of the study could contribute in the development of guidelines to prevent infertility or to nutritional management associated to infertility treatments to improve reproductive performance. Furthermore, the elucidation of the role of adiponectin and follistatin in female reproductive functions and its association with dietary variables and the IVF outcomes could lead to the use of adiponectin or follistatin as therapeutic targets in novel treatment strategies of infertility disorders.

ELIGIBILITY:
Inclusion Criteria:

* Presence of subfertility (male or female origin)

Exclusion Criteria:

* Women's age <41.
* Previous IVF attempt or pregnancy.
* Female obesity (BMI>30 kgr/m2).
* Endometriosis
* Oocyte donation.
* Adherence to a hypocaloric diet for weight loss or changes in dietary habits during the last six months.
* Presence of female diabetes mellitus, cardiovascular disease, hypertension, neoplasm, hypothyroidism or psychiatric disorders.
* Previous ovarian surgery.
* Natural cycle IVF.
* Couples whose male partner shows an abnormality of the male genital tractus : Varicocele, undescended testis, testicular volume < 12ml

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subfertile couples undergoing IVF treatment at a Fertility Clinic in Athens
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Live Birth | 9 months
  Birth of a neonate on or after 24 weeks gestation

SECONDARY OUTCOMES:
Hormonal profile | 3 months
  Baseline serum E2, anti-mullerian hormone, inhibin b, luteinizing hormone, follicle stimulating hormone concentrations.
Oocyte number. | 3 months
  Total Number of oocytes produced.
Oocyte quality. | 3 months
  The morphological feature of each oocyte wil be evaluated with the aid of inverted microscope. The criteria employed for the morphological evaluation of oocytes are: a. normal oocytes showed clear cytoplasm with homogenous fine granularity; b. granular oocytes, dark with granularity either homogenous in whole cytoplasm or concentrated in the central portion of oocyte; c. cytoplasmic inclusions comprised vacuoles presumed to be of endocytotic origin; d. anomalies of zona pellucida e. fragmented polar body of different sizes; f. non-spherical shape of oocyte; and g. wide perivitelline space.
Embryo number. | 3 months
  Total Number of embryos produced.
Embryo quality. | 3 months
  Embryo morphology will be assessed as follows: 44 h ± 1 h after intracytoplasmatic sperm injection, for day two evaluation and 68h ± 1 h after intracytoplasmatic sperm injection, for day 3 evaluation. Embryo morphology will be carried out using an inverted microscope
Semen volume. | 1 month.
  Ejaculate volumes will be estimated by specimen weight, assuming a semen density of 1.0 g/ml.
Semen concentration. | 1 month.
  Sperm concentration will be evaluated by hemocytometer Motility will be assessed in accordance with the World Health Organization 2010 criteria
Semen morphology. | 1 month.
  Regarding semen morphology, the World Health Organization criteria as described in 2010 state that a sample is normal if 4% (or 5th centile) or more of the observed sperm have normal morphology.
Semen Motility. | 1 month.
  Motility will be assessed in accordance with the World Health Organization 2010 criteria and classified as progressive motile (A + B), total motile (A + B + C), or immotile (D).
Fertilization rate | 3 months
  Fertilization rate will be determined on day 1 after the IVF/intracytoplasmatic sperm injection procedure, and is going to calculated as the number of fertilized oocytes divided by the total number of oocytes retrieved
Serum Adiponectin | 6 months
  Serum adiponectin levels will be measured by ELISA method on day 1 of the ovarian stimulation protocol, on day 3, on day 5, on day 7, on day 9 and the day of oocyte retrieval.
Follicular Fluid Adiponectin | 6 months
  Follicular fluid adiponectin levels from the dominant oocyte will be measured by ELISA method.
Follicular Fluid Follistatin, | 6 months
  Follicular fluid follistatin levels from the dominant oocyte will be measured by ELISA method.
Clinical Pregnancy | 6 months
  Elevation in b-human chorionic gonadotropin with the confirmation of an intrauterine pregnancy by ultrasound, first performed at 6 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Yiannakouris, PhD, Principal Investigator — Associate Professor of Physiology
Locations (1):
- Harokopio University, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karayiannis D, Kontogianni MD, Mendorou C, Douka L, Mastrominas M, Yiannakouris N. Association between adherence to the Mediterranean diet and semen quality parameters in male partners of couples attempting fertility. Hum Reprod. 2017 Jan;32(1):215-222. doi: 10.1093/humrep/dew288. Epub 2016 Nov 14. PMID 27994040
- [Derived] Karayiannis D, Kontogianni MD, Mendorou C, Mastrominas M, Yiannakouris N. Adherence to the Mediterranean diet and IVF success rate among non-obese women attempting fertility. Hum Reprod. 2018 Mar 1;33(3):494-502. doi: 10.1093/humrep/dey003. PMID 29390148